CLINICAL TRIAL: NCT02805829
Title: Combination Trastuzumab With Expanded NK Cells for Treating HER2-positive Gastric Cancer
Brief Title: Combination Trastuzumab With Expanded Natural Killer Cells for Treating HER2-positive Gastric Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Junnian Zheng, professor, Xuzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2016-KL014-01
Record Dates: First submitted 2016-06-15; First posted 2016-06-20 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Gastric Cancer
Keywords: NK cells; Trastuzumab
MeSH Terms: conditions — Stomach Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Trastuzumab + NK cells (Experimental): On Cycle 1,day -2, patients will receive IV loading dose 8mg/Kg trastuzumab, followed by collection blood on day 0. After NK expansion and verification that the resulting NK cells meet release criteria, NK cells were washed and resuspended in isotonic sodium chloride for intravenous transfusion on day 14.
  NK cellular therapy conduct 2 cycles per year. The maintenance dose of trastuzumab monotherapy is 6 mg/kg over 30 to 90 minutes IV infusion every 3 weeks till to disease progress.
  Interventions: Drug: Trastuzumab + NK cells

INTERVENTIONS:
Drug: Trastuzumab + NK cells — NK cellular therapy conduct 2 cycles per year. Herceptin initial dose of 8 mg/kg over 90 minutes IV infusion, followed by 6 mg/kg over 30 to 90 minutes IV infusion every 3 weeks till to disease progress.
  Other Names: Herceptin

SUMMARY:
This trial is to evaluate the safety and effectiveness of activated and expanded in vitro autologous NK cells following trastuzumab treatment for patients Human Epidermal Receptor-2 overexpressing advanced gastric cancer.

DETAILED DESCRIPTION:
Tumor antigen-specific monoclonal antibodies, block oncogenic signaling and induce Fcγ receptor (FcγR)-mediated cytotoxicity, are considered to be one of the most successful strategies in cancer therapy. Trastuzumab, a monoclonal antibody directed against HER2, was investigated in combination with chemotherapy for first-line treatment of HER2-positive advanced gastric cancer. The use of cellular immunotherapy has increased significantly over the past two decades. Natural killer cells are lymphocytes of the innate immune system that have the ability to recognize and kill malignant cells. There is growing evidence show antibody-dependent cell-mediated cytotoxicity (ADCC) by NK cells contributes to the efficacy of Herceptin. Therefore, methods to enhance ADCC, such as stimulating the innate immune response, may clinically translate to improved antitumor activity. In this study, the investigators sought to enhance the clinical activity of trastuzumab, administrated in combination with expanded autologous NK cells. The enrolled patients are diagnosed HER2+ advanced gastric cancer. The eligible patient will administrate herceptin on 2 days prior to blood collection. The initial dose of herceptin is 8 mg/kg over 90 minutes IV infusion. On day 0 peripheral blood mononuclear cells were separated from 40-50ml blood by density gradient centrifugation. Then were cultured with human NK cell culture medium and stimulation cytokines in a humidified, 5% carbon dioxide incubator for about 14 days. After NK expansion and verification that the resulting NK cells meet purity, gram stain, and endotoxin release criteria, NK cells were washed and resuspended in isotonic sodium chloride. NK cellular therapy conduct 2 cycles per year. The maintenance dose of herceptin monotherapy is 6 mg/kg over 30 to 90 minutes IV infusion every 3 weeks. This study will determine the safety and efficacy of this novel combinational therapeutic strategy in HER2 positive gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to 18 years or older;
* Patients with histologically confirmed HER2 positive advanced gastric cancer through immunohistochemistry (IHC) and fluorescence in situ hybridization (FISH);
* Normal marrow hematopoiesis function: Hemoglobin≥90g/L, White Blood Cell count≥4000/μL, absolute Neutrophil Cell count (ANC)≥1500/μL, Platelet≥100000/μL;
* Normal important organ function: Total bilirubin≤1.5-fold institutional upper limit of normal (ULN), Aspartate aminotransferase and Alanine aminotransferase≤2.5-fold ULN, Creatinine clearance≥80mL/min;
* Life expectancy≥6 months;
* No other serious heart, lung, kidney dysfunction;
* Quality of life (Karnofsky performance score)≥60;
* Patient must be able to understand and be willing to sign a written informed consent document.

Exclusion Criteria:

* Prior allergic reaction or hypersensitivity to cytokines (eg.Interleukin-2);
* Patients with systemic or local infection requiring anti-infections treatment;
* Patients currently treated with systemic immunosuppressive agents, including steroids;
* Patients with active autoimmune disease or history of transplantation requiring steroid treatment;
* Tested positive for HIV;
* Pregnant or lactating women;
* Patients with coagulation disorders;
* Patients with important organ dysfunction, including cardiac, lung, liver;
* Patients experiencing a cardiac events (acute coronary syndrome, myocardial infarction or ischemia) within the 3 months;
* Any reason that, in the opinion of the investigator, contraindicates that the patient participates in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-01; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 2 years

SECONDARY OUTCOMES:
Number of Participants with tumor recurrence metastasis as a Measure of effectiveness | 2 years

OTHER OUTCOMES:
T cell subsets figures | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Junnian Zheng, MD, Principal Investigator — Xuzhou Medical University
Locations (1):
- Xuzhou medical university, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No